CLINICAL TRIAL: NCT04560855
Title: Secure Self-monitoring Through a Combination of Connected Objects: Implementation in COVID-19 Patients Monitored at Home
Acronym: SECURADOM
Status: Completed | Type: Observational
Sponsor: Withings (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-A00981-38
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2020-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid19 Patients: Patients diagnosed as COVID-19 positive and managed on an outpatient basis.
  Interventions: Device: Connected devices measurements

INTERVENTIONS:
Device: Connected devices measurements — The patient has to measure everyday several vital parameters like respiration and heart rate during the night with Withings Sleep, temperature with Withings Thermo, arterial pressure with Withings Tensiometer and physical activity with Withings smartwatch.

SUMMARY:
Currently, COVID+ infected patients who are on ambulatory home monitoring self-assess their health status simply by completing questionnaires and measuring their temperature twice a day. The SECURADOM project proposes to facilitate the follow-up of COVID+ or suspected COVID+ infected patients, followed at home, by collecting clinical signs on a telephone application and to monitor physiological safety parameters (respiratory rate, heart rate, temperature, blood pressure, activity) using connected objects developed by the company WITHINGS. This daily monitoring, which can be transmitted by patients to the doctors in charge of their surveillance, will improve the quality and safety of home monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adults, men and women, 18 y/o or more
* Patient diagnosed COVID positive with RT-PCR positive or very suggestive symptoms and a contagion (contact with sick subjects) that can be managed on an outpatient basis.
* Patient in possession of a smartphone (with Android or iOS) allowing the installation of the Withings Health Mate application
* Patient with access to an internet connection for the use of Withings connected products at the containment site
* Voluntary patient who has not objected to his or her participation
* Patient affiliated to or beneficiary of a social security scheme

Exclusion Criteria:

* Pregnant Women
* Patient with severe symptoms requiring hospitalization as recommended by the French Ministry of Health (23/03/2020)
* Patient without social protection or affiliated to the AME (State Medical Aid)
* Person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure (patient under guardianship or curatorship) Articles L1121-5 to L1121-8
* Patient who, in the judgment of the investigator, may not be cooperative or respectful of the obligations inherent to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed COVID positive with RT-PCR positive or very suggestive symptoms and a contagion (contact with sick subjects) that can be managed on an outpatient basis.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the patient's aggravation with a logistic regression model | 1 year
  The sensitivity and specificity of a logistic regression model based on the vital parameters retrieved from the connected devices will be calculated in order to evaluate its performance
Sensitivity and Specificity of the patient's aggravation with a cluster model | 1 year
  The sensitivity and specificity of a cluster model based on the vital parameters retrieved from the connected devices will be calculated in order to evaluate its performance

SECONDARY OUTCOMES:
Study the evolution of daily patient parameters without aggravation over time | 1 year
  Slope of daily patient parameters without aggravation over time.
Subjective assessment of the connected devices | 1 year
  The UX meCUE Scale (User eXperience modular evaluation of key Components of User Experience) questionnaire will be used. It is composed of 16 items where the participant has to answer if he agrees or not with the statement (from 0 - don't agree - to 6 - strongly agree -).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pépin, Pr, Principal Investigator — CHU Grenoble Alpes
Locations (4):
- France (4):
  - CHU Grenoble-Alpes, Grenoble, Auvergne-Rhône-Alpes
  - CHU d'Amiens, Amiens, Hauts-de-France
  - Hôpital d'Instruction des Armées Percy, Clamart, Île-de-France Region
  - Hôpital d'Instruction des Armées Bégin, Saint-Mandé, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No